CLINICAL TRIAL: NCT01347047
Title: Institutional Registry of Amyloidosis (Hospital Italiano de Buenos Aires)
Brief Title: HIBA-Institutional Registry of Amyloidosis
Acronym: RIA-HIBA
Status: Recruiting | Type: Observational
Sponsor: Hospital Italiano de Buenos Aires (Other)
Collaborators: Instituto Cardiovascular de Buenos Aires (Other); Austral University, Argentina (Other); Hospital de Alta Complejidad en Red (Other); Hospital de Clinicas José de San Martín (Other); HOSPITAL BRITANICO DE BUENOS AIRES (Other); Hospital Privado de Rosario (Unknown); Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other); La Fundacion Favaloro para la Investigacion y la Docencia Medica (Other); Sanatorio Anchorena (Unknown); Centro Médico Uruguayo, Uruguay (Unknown); Clínica Foianini, Bolivia (Unknown)
Responsible Party: Principal Investigator, MARIA LOURDES POSADAS MARTINEZ, MD, PHD, Hospital Italiano de Buenos Aires
Other Study IDs: 1675
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Amyloidosis
Keywords: Amyloidosis; Known or Suspected; rare diseases
MeSH Terms: conditions — Amyloidosis; Rare Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Creating a population-based registry system Amyloidosis prospective epidemiological survey

   * risk factors
   * diagnosis
   * prognosis
   * treatment
   * monitoring
   * survival
2. Describe the occurrence of amyloidosis in the population of HIBA, Hospital Italiano de Buenos Aires.
3. Describe the characteristics of clinical presentation, evolution and predisposing factors of amyloidosis.

DETAILED DESCRIPTION:
Amyloidosis is a systemic disease that is usually a result of misfolded proteins in the form of amorphous fibrillar material in various tissues and can cause progressive dysfunction of the same. The prevalence of amyloidosis varies depending on the population concerned and the type of amyloid. While prevalence in the general population is unknown, according to estimates by the Mayo Clinic this prevalence is 1 in 90 666% in the U.S. In England this disease generated about 0.0084% (1367 / 16232579) of all hospital visits between April 2008 and April 2009.

The most common clinical manifestations include cardiac disease, renal and liver function, but it may vary widely depending on the type of amyloidosis, the organ infected and extent of the deposits. Amyloid infiltration can produce signs and symptoms that may be very similar to other rheumatic diseases. This may suggest potential clinical polymorphic underdiagnosis due to low clinical suspicion.

The registries are organized systems of systematic data collection of a large number of patients quickly and efficiently on a particular disease at a given time.

The main difficulty of the registries is the guarantee of the quality of their data.

The main objectives of the registry are:

1. Understand risk factors and prognosis.
2. Evaluate the diagnostic and therapeutic comparison with current standards.
3. Advance knowledge of the disease to optimize the assessment, treatment and monitoring of patients.
4. Analyze the effectiveness of new therapies.
5. Studying differences between populations.
6. Quickly estimate the morbidity, mortality and resource utilization associated with a disease entity.
7. Examine the course of a disease
8. Formulate novel hypotheses for further prospective studies. Currently, there are registries for patients with transthyretin amyloidosis (TAHOS), global registry of transplant patients with familial amyloid poly neuropathy. Also, there are indirect registries such as the kidney transplant, heart transplant, among others.

The investigators found no data on the prevalence or incidence, evolution and prognosis of amyloidosis in our country. There are no existing records of national Amyloidosis in Latin America that could describe the behavior of this disease in our environment. Because it is a chronic disease with amyloid infiltration and can produce signs and symptoms that may be very similar to other rheumatic diseases, this clinic potentially poliform, may suggest underestimation of low clinical suspicion. As there is no cure, some patients may persist symptomatic despite adequate therapy, that is why it is important the creation of a monitoring system to generate data on the evolution and prognosis. The data registries can be used to develop new treatment guidelines and recommendations, also to inform and educate physicians on the management of this disease.

The Hospital Italiano de Buenos Aires is a center of high complexity of derivation of this type of pathology and due to the fact that the hospital, that has a private health insurance system (HIBA's health plan [plan de salud, PS], gives the unique opportunity denominators for the generation of a population on their affiliates, therefore the investigators propose to make a Institutional Registry of Amyloidosis.

ELIGIBILITY:
Cases of amyloidosis are captured by electronic medical records whenever the physician register amyloidosis as a patient diagnosis, and/or there is amyloidosis in a biopsy specimen and/or requests for the following studies of an adult patient: plasma kappa and lambda light-chain concentrations, the kappa: lambda ratio, transthoracic Doppler echocardiography, or cardiovascular magnetic resonance examination or pyrophosphate scintigraphy From the possible cases included in the IRA, a prospective review of the electronics health records was performed to confirm the presence of amyloidosis

**Inclusion Criteria: 1 AND (2 or 3)

1. Patients over 18 years:
2. Confirmed amyloidosis: Proof of deposit of amyloid pathology by tissue biopsy in abdominal fat, bone marrow, rectum or organ involved (eg, kidney, liver, sural nerve)
3. Clinically compatible case of Amyloidosis :

   * Exclusion Criteria:

Refusal to participate in the study or the informed consent process by the patient or legal representative or refusal to consent to participate in the study in the case of minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over 18 years old with diagnosis or suspected amyloidosis of Italiano Hospital of Buenos Aires
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-04 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Epidemiologic characteristics | From inclusion date (daignosis) until the date of death from any cause or date of last follow up(if not dead) assessed up to 10 years
  Survival anual
Epidemiologic characteristics | From treatment date until the date of best organ response or documented progression or date of death from any cause, whichever came first, assessed up to 10 years
  Organ response
From treatment to folow up, annualy | at baseline
  Baseline description
Treatment patterns | From diagnosis, evaluated after every line of treatment or annualy up to 10 years
  Type of treatment, duration, adverse events, completition

CONTACTS AND LOCATIONS:
Overall Officials: María Lourdes Posadas-Martínez, MD, Principal Investigator — Hospital Italiano de Buenos Aires, Argentina; Elsa Nucifora, MD, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Diego Hernan Giunta, MD, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Dorotea Fantl, MD, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Gustavo Greloni, MD, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Maria Adela Aguirre, MD, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Cesar Antonio Belziti, MD, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Patricia Sorroche, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Soledad Saez, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Erika Brulc, MD, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Diego Perez de Arenaza, MD, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Eugenia Villanueva, MD, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Marcelina Carretero, MD, Study Chair — Hospital Italiano de Buenos Aires, Argentina; Carolina María Petit Cwirko, MD, Principal Investigator — Clinica Foianini, Santa Cruz, Bolivia; Pablo Young, MD, Principal Investigator — Hospital Británico, Buenos Aires, Argentina; Gisela Streitenberger, MD, Principal Investigator — Hospital de Alta Complejidad El Cruce Nestor Kirchner, Buenos Aires, Argentina; Luciana Leon Cejas, MD, Study Chair — Hospital Británico, Buenos Aires, Argentina; Veronica Volberg, MD, Principal Investigator — Hospital de Clínicas José de San Martin, Buenos Aires, Argentina; Sergio Juan Baratta, MD, Principal Investigator — Hospital Austral, Buenos Aires, Argentina; Juan Pablo Costabel, MD, Principal Investigator — Instituto cardiovascular Buenos Aires, Argentina; Carlos Dumont Dunayevich, MD, Principal Investigator — Hospital Privado de Rosario, Santa Fe, Argentina; Alejandro Quiroga, MD, Principal Investigator — Fundación Favaloro, Buenos Aires, Argentina; Adrian Fernandez, MD, Study Chair — Fundación Favaloro, Buenos Aires, Argentina; Josefina Parodi, MD, Principal Investigator — Anchorena, Buenos Aires, Argentina; Franco Leoni, MD, Study Director — Médica Uruguaya, Uruguay; Eduardo Ortuño Campos, MD, Study Director — Hospital Universitarios Austral, Buenos Aires, Argentina; Jorge Thierer, MD, Principal Investigator — CEMIC, , Buenos Aires, Argentina
Locations (1):
- Hospital Italiano de Buenos Aires, Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT01347047/Prot_SAP_000.pdf